CLINICAL TRIAL: NCT05682638
Title: A Global Multi-center, Randomized, Blinded, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine for the Prevention of COVID-19 in Participants Aged 18 Years and Older
Brief Title: A Global Multi-center Clinical Study of SARS-CoV-2 mRNA Vaccine for the Prevention of COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: AIM Innovation Biotechnology (Shanghai) Co., Ltd (Unknown); Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry); LiveRNA Therapeutics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LVRNA009-II/III-01
Record Dates: First submitted 2023-01-08; First posted 2023-01-12 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2
Keywords: mRNA, Prevention
MeSH Terms: interventions — LVRNA009 COVID-19 vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine group (Experimental): Phase 3(Base the result of Phase 1 and Phase 2, intervent 100μg): initial vaccination stage- LVRNA009; crossover vaccination stage- placebo
  Interventions: Biological: LVRNA009; Other: 0.9%NaCl
- Control group (Placebo Comparator): Phase 3: initial vaccination stage- placebo; crossover vaccination stage- LVRNA009
  Interventions: Biological: LVRNA009; Other: 0.9%NaCl

INTERVENTIONS:
Biological: LVRNA009 — 100μg/1.0ml/dose(50 μg/0.5ml/Vial), 2 injection with 28 days apart
Other: 0.9%NaCl — 1.0ml/dose, 2 injection with 28 days apart

SUMMARY:
A Global Multi-center, Randomized, Blinded, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (LVRNA009) for the Prevention of COVID-19 in Participants Aged 18 Years and Older

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older.
2. Understand the content of the Informed Consent Form (ICF), and voluntarily sign the ICF (If the participant is unable to sign the ICF on his/her own due to illiteracy, an impartial witness is needed).
3. Participants who are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.
4. Female participants of childbearing potential or partners of male participants:

   voluntarily agree to use effective contraception with their partners prior to the first vaccination and must agree to continue such precautions during the study until 3 months after full vaccination (including the initial set of vaccination and crossover set of vaccination). [Effective contraception includes oral contraceptives, injectable or implantable contraception, extended-release topical contraceptives, hormonal patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (for male), diaphragms, cervical caps, etc.].
5. For female participants: without childbearing potential (amenorrhea for at least 1 year or documented surgical sterilization) or have used effective contraception with a negative pregnancy test before each vaccination in this study.
6. On the day of 1st dose of vaccination and 24 hours prior to vaccination, axillary temperatures <37.3°C/99.1°F.
7. Healthy participants or participants with mild underlying disease [in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study].

Exclusion Criteria:

1. History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS), or other coronavirus infections.
2. Individuals using prescription medications for prophylaxis or treatment of SARS-CoV-2 (including vaccination of licensed COVID-19 vaccines).
3. History of a previous laboratory-confirmed diagnosis of SARS-CoV-2 infection or COVID-19.
4. History of allergy to any component of the study vaccine or history of severe allergic reaction to vaccine or drug (including but not limited to anaphylaxis, allergic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, or localized allergic necrosis (Arthus reaction)).
5. Positive nucleic acid for SARS-CoV-2 in nasopharyngeal/oropharyngeal swab specimens.
6. Positive HIV test results.
7. A history or family history of convulsions, epilepsy, encephalopathy and psychosis.
8. Malignant tumors in the active phase, malignant tumors not receiving adequate treatment, malignant tumors at potential risk of recurrence during the study period.
9. Asplenia or functional asplenia, complete or partial splenectomy from any cause.
10. Prolonged (defined as more than 14 days) use of immunosuppressive or other immunomodulatory drugs (e.g., corticosteroids, ≥20 mg/d prednisone or equivalent; however, inhaled and topical steroids are permitted) within 6 months prior to the 1st dose of investigational vaccine.
11. Any other licensed vaccines given within 28 days prior to the study vaccination, or planned administration of vaccine(s) within 28 days after the 2nd dose in the blinded crossover vaccination.
12. Have received immunoglobulin or other blood products within 3 months prior to enrollment or plan to receive them during the study period.
13. Blood donation or blood loss ≥ 450 mL within 1 month prior to enrollment or planned to donate blood during the study period.
14. Participants who have received any other investigational product within 1 month prior to enrollment or intent to participate in another clinical study at any time during the conduct of this study.
15. Women who are pregnant or breastfeeding.
16. Participants deemed unsuitable for participation in this study based on the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34000 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring in SARS-CoV-2 naive participants in vaccine(100μg) group | From 14 days after the 2nd dose in the initial set of vaccination

SECONDARY OUTCOMES:
The person-year incidence density of first episodes of virologically-confirmed moderate to severe cases of COVID-19 for SARS-CoV-2 naive participants | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed severe cases of COVID-19 for SARS-CoV-2 naive participants | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 leading to death for SARS-CoV-2 naive participants | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring for SARS-CoV-2 naive participants at different age strata (18-59 years, ≥60 years) | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring for SARS-CoV-2 non-naive participants | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed severe cases of COVID-19 for SARS-CoV-2 non-naive participants | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring regardless prior SARS-CoV-2 infection | From 14 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring | From the 1st dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring | From 7 days after the 2nd dose in the initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed moderate to severe cases of COVID-19 for SARS-CoV-2 native participants | From 14 days after the 2nd dose in the crossover set of vaccination
The person-year incidence density of first episodes of virologically-confirmed severe cases of COVID-19 for SARS-CoV-2 naive participants | From 14 days after the 2nd dose in the crossover set of vaccination
The person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 leading to death regardless prior SARS-CoV-2 infection | From 14 days after the 2nd dose in the crossover set of vaccination
Incidence, severity and duration of each solicited (local and systemic) Adverse Event (AE) | Within 14 days post each dose in reactogenicity subgroup in the initial set of vaccination
Incidence, severity, and causality of AEs occurring | 0-28 days post each dose
Incidence, severity, and causality of Serious Adverse Events (SAEs) | From the day of 1st dose in the initial set of vaccination to 12 months after the 2nd dose in crossover set of vaccination
Incidence, severity, and causality of Adverse Events of Special Interest (AESIs) | From the day of 1st dose in the initial set of vaccination to 12 months after the 2nd dose in crossover set of vaccination
Incidence, severity, and causality of pregnancy events | From the day of 1st dose in the initial set of vaccination to 12 months after the 2nd dose in crossover set of vaccination
Geometric mean Titer (GMT) of SARS-CoV-2 virus neutralizing antibody responses and S-protein IgG antibody responses of the initial set of vaccination or the day of crossover vaccination (whichever comes earlier) | 14 days, 28 days, 3 months and 6 months after the 2nd dose
Geometric mean Titer (GMT) of SARS-CoV-2 virus neutralizing antibody responses and S-protein IgG antibody responses in the crossover set of vaccination | 28 days, 3 months, 6 months and 12 months after the 2nd dose
Geometric mean Increase (GMI) of SARS-CoV-2 virus neutralizing antibody responses and S-protein IgG antibody responses of the initial set of vaccination or the day of crossover vaccination (whichever comes earlier) | 14 days, 28 days, 3 months and 6 months after the 2nd dose
Geometric mean Increase (GMI) of SARS-CoV-2 virus neutralizing antibody responses and S-protein IgG antibody responses in the crossover set of vaccination | 28 days, 3 months, 6 months and 12 months after the 2nd dose
The seroconversion rate (SCR) of SARS-CoV-2 virus neutralizing antibody and S-protein IgG antibodies in seronegative participants at baseline of the initial set of vaccination or the day of crossover vaccination (whichever comes earlier) | 14 days, 28 days, 3 months and 6 months after the 2nd dose
The seroconversion rate (SCR) of SARS-CoV-2 virus neutralizing antibody and S-protein IgG antibodies in seronegative participants at baseline in the crossover set of vaccination | 28 days, 3 months, 6 months and 12 months after the 2nd dose
The seroconversion rate (SCR) of SARS-CoV-2 virus neutralizing antibody and S-protein IgG antibodies in seropositive participants at baseline of the initial set of vaccination or the day of crossover vaccination (whichever comes earlier) | 14 days, 28 days, 3 months and 6 months after the 2nd dose
The seroconversion rate (SCR) of SARS-CoV-2 virus neutralizing antibody and S-protein IgG antibodies in seropositive participants at baseline in the crossover set of vaccination | 28 days, 3 months, 6 months and 12 months after the 2nd dose

OTHER OUTCOMES:
Cellular immune subgroup: The specific cellular immune response (IL-2) to SARS-CoV-2 (ELISpot) | 7 days, 14 days, 28 days after the 2nd dose of the initial set of vaccination
Cellular immune subgroup: The specific cellular immune response (IL-4) to SARS-CoV-2 (ELISpot) | 7 days, 14 days, 28 days after the 2nd dose of the initial set of vaccination
Cellular immune subgroup: The specific cellular immune response (IL-13) to SARS-CoV-2 (ELISpot) | 7 days, 14 days, 28 days after the 2nd dose of the initial set of vaccination
Cellular immune subgroup: The specific cellular immune response (IFN-γ) to SARS-CoV-2 (ELISpot) | 7 days, 14 days, 28 days after the 2nd dose of the initial set of vaccination
Cross-neutralization subgroup: The cross-neutralizing ability of serum neutralizing antibodies | 14 days and 28 days after the 2nd dose of the initial set of vaccination
The immunological correlation of risk and protection against symptomatic COVID-19 and SARS-CoV-2 infection | 6 months after initial set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring for SARS-CoV-2 naive participants | From 14 days after the 2nd dose in the crossover set of vaccination
The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring for SARS-CoV-2 non-naive participants | From 14 days after the 2nd dose in the crossover set of vaccination
The person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 of any severity occurring caused by individual Variants of Concern (VOCs) | From 14 days after the 2nd dose in the initial set of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI CRDR Research Annex, Siaya Country Referral Hospital, Siaya, Kenya